CLINICAL TRIAL: NCT00228332
Title: A Double-Blind, Placebo-Controlled Trial Investigating the Effect of a Treatment With Zinkgluconaat for Verrucae Vulgares
Brief Title: A Trial Investigating the Effect of a Treatment With Zinkgluconaat for Verrucae Vulgares
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2004/005
Record Dates: First submitted 2005-09-13; First posted 2005-09-28 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Verrucae Vulgares

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Administration of zinkgluconaat or placebo

SUMMARY:
A Double-blind, placebo-controlled trial investigating the effect of a treatment with zinkgluconaat for verrucae vulgares

DETAILED DESCRIPTION:
A Double-blind, placebo-controlled trial investigating the effect of a treatment with zinkgluconaat for verrucae vulgares

ELIGIBILITY:
Inclusion Criteria:

* Patients with verrucae vulgares

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2004-04; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Disappearence of the verrucae vulgares after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Annelies Stockman, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be